CLINICAL TRIAL: NCT02881294
Title: A Phase I, Single-center, Open-label, Single-dose Study to Evaluate the Effect of Food, Gender, and Age on the Pharmacokinetic Profile of Orally Administered SUVN-G3031 in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Food, Gender, and Age on the Pharmacokinetic Profile of SUVN-G3031 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP1S23031H3
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction | interventions — samelisant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Food Effect (Active Comparator): SUVN-G3031 tablets single dose
  Interventions: Drug: SUVN-G3031
- Gender Effect (Active Comparator): SUVN-G3031 tablets single dose
  Interventions: Drug: SUVN-G3031
- Age Effect (Active Comparator): SUVN-G3031 tablets single dose
  Interventions: Drug: SUVN-G3031

INTERVENTIONS:
Drug: SUVN-G3031

SUMMARY:
The purpose of the study is to investigate the effect of Food, Gender, and Age on the Pharmacokinetic Profile of SUVN-G3031 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18 to 45 years with a BMI between 18 and 30 kg/m2, (inclusive) for food and gender effect
* Healthy male aged 60 to 70 years with a BMI between 18 and 32 kg/m2, (inclusive) for age effect

Exclusion Criteria:

* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs as judged by Investigator.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the study drug.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody
* History of any important clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Area under concentration (AUC) | 96 hours
Maximum observed concentration (Cmax) | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles, Overland Park, Kansas, United States